CLINICAL TRIAL: NCT00049959
Title: A Randomized, Placebo-Controlled, Masked, Multicenter Phase III Study Of Photodynamic Therapy With Verteporfin For Injection (VFI) For The Treatment Of Multiple Basal Cell Carcinoma
Brief Title: Two Studies to Determine if Verteporfin PDT is Effective & Safe in Treating Multiple Basal Cell Carcinoma of the Skin.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VFI MBCC 01 and VFI MBCC 02
Record Dates: First submitted 2002-11-15; First posted 2002-11-19 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-03

CONDITIONS: Basal Cell Carcinoma; Nevoid Basal Cell Carcinoma Syndrome; Gorlin Syndrome
Keywords: Verteporfin PDT; multiple basal cell carcinoma; nevoid basal cell carcinoma syndrome
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome; Basal cell carcinoma, multiple

INTERVENTIONS:
Drug: verteporfin PDT

SUMMARY:
The purpose of the two studies is to determine whether an experimental therapy using a photoactive drug, verteporfin, in combination with direct light exposure of basal cell carcinoma of the skin can safely eliminate these skin tumors.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) of the skin is the most common type of cancer that can be treated with various therapies including surgical removal. A number of factors can lead to the development of multiple BCC of the skin, including genetic disorders (e.g., nevoid basal cell carcinoma syndrome). Treatment of multiple BCC becomes much more challenging. In these trials, the experimental therapy: verteporfin PDT is compared to placebo PDT. PDT or photodynamic therapy in these studies is the combination of the photoactive drug verteporfin (given intravenously) and red light exposure of skin tumors.

The primary objective is to assess whether verteporfin PDT can completely eliminate multiple BCCs. Eligible subjects will have at least 3 BCCs. Study subjects won't know which treatment they have been been assigned to - this is done randomly (like flipping a coin). After study treatment, the BCCs in each subject will be closely observed and toward the end of the study all will be surgically removed and examined to verify response to study treatment. Safety will be assessed by testing blood samples before and after study treatment, and analyzing adverse events and skin reactions to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Currently has at least 3 eligible BCC skin tumors that have never been treated
* Is willing to have these tumor sites surgically removed

Exclusion Criteria:

* Has xeroderma pigmentosum
* Has BCC tumors that are the result of prior radiotherapy or immunosuppression due to an organ transplant
* Is immunosuppressed
* Has abnormal liver function
* Is receiving systemic chemotherapy or has received chemotherapy within the last two years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herma Neyndorff, Study Director — QLT Inc.